CLINICAL TRIAL: NCT03762863
Title: Retention of Tourniquet Application Skills Following Participation in a Bleeding Control Course
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Somerville Office of Emergency Management (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QMREC2206a
Record Dates: First submitted 2018-11-29; First posted 2018-12-04 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Hemorrhage
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Appropriate application of a CAT tourniquet (Experimental): All study subjects attended an American College of Surgeons Stop the Bleed Basic course with live training by approved instructors. 6 months after participation in the Stop the Bleed class volunteers study subjects are randomly solicited to return for a refresher session. During this refresher session the volunteer study subjects are observed to determine if they have retained tourniquet application skills and to what degree they have retained them. A 10 point check list will be used to evaluated tourniquet application skill retention.
  Interventions: Device: Tourniquet application skill retention

INTERVENTIONS:
Device: Tourniquet application skill retention — Tourniquet application following the procedure as learned in the Stop the Bleed curriculum.
  Other Names: Evaluation of retention of critical steps in tourniquet application 6 months after attending a Stop the Bleed class.

SUMMARY:
Prospective, observational study of students 6 months after completing a Stop the Bleed course to determine overall ability to effectively use a tourniquet to stop external extremity hemorrhage. Following the release of the Hartford Consensus in October 2015, the American College of Surgeons Committee on Trauma initiated the National Stop the Bleed campaign (2) that among several proactive recommendations was to encourage first responders and the lay public to become trained, equipped and empowered to step forward and intervene in a bleeding emergency. The Stop the Bleed initiative provides baseline education and training in the use of tourniquets to stop extremity hemorrhage when pressure alone does not work. While the program has progressively provided education and training to over 130,000 individuals worldwide there are no recommendations regarding time intervals for refresher training to maintain confidence and competence in the use of tourniquets. The rationale for this study is to ascertain if tourniquet application skills are sufficiently maintained 6 months after participation in a Stop the Bleed course and to provide recommendations for refresher training based on the results.

DETAILED DESCRIPTION:
In response to an alarming rise in active shooter/hostile incidents in the United States, in 2013 the American College of Surgeons convened a committee of multidisciplinary trauma experts who in collaboration with the federal government created a protocol for a national policy to enhance survivability from these active shooter incidents as well as other intentional mass casualty events. The committee's recommendations were called the Hartford Consensus. Among the recommendations of the Hartford Consensus was the training of first responders (law enforcement, EMS and fire personnel) as well as the public (so-called "immediate responders") in the basics of bleeding control. In October 2015, responding aforementioned recommendation, the White House launched the Stop the Bleed national awareness campaign as a "call to action". Under the auspices of the American College of Surgeons Committee on Trauma, a curriculum was developed teaching responders how to recognize and intervene in the event of catastrophic bleeding. Of the three bleeding control interventions promoted (external pressure, wound packing and tourniquet application) the tourniquet application component of the Stop the Bleed curriculum is evidence-based and provides the student with both didactic and psychomotor education. To date there is a paucity of data available to provide insight as to how long this vital skill is retained. More over there is no recommendation on refresher education with additional opportunities to practice this life-saving procedure. This study will serve as a follow-up to Stop the Bleed (also called Bleeding Control or B-Con) education provided by the investigator. The intent is to bring participants from a Bleeding Control course back to the investigator 6 months following initial education and assess their retention of tourniquet application skills. All participants will be assessed using a tourniquet simulator and their success will be measured in their ability to stop the bleeding using the simulator. The participants will be observed for proper identification of bleeding necessitating the use of a tourniquet, selection of the proper site of application, proper application of the device (use as described in the Stop the Bleed curriculum). This study will not involve the use of actual patients or human subjects. It is intended to be follow up assessment to skills-based education with an endpoint that will provide insight as to a time-frame for refresher training. Of the three bleeding control skills taught as part of the Stop the Bleed curriculum, the application the tourniquet is a universal stop the bleed intervention and most likely intervention to be used to stop the bleed.

ELIGIBILITY:
Inclusion Criteria:

All adults (18 years of age and above) participating in an American College of Surgeons Sponsored "Stop the Bleed" course

Exclusion Criteria:

1. Less than 18 years of age
2. Any participant that attends another program that includes tourniquet application skills after attendance at the Stop the Bleed program
3. Any participant that does not consent for inclusion for study data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Tourniquet application retention | 6 months
  A 10 point data collection checklist was developed paralleling the procedure for tourniquet application as set forth in the American College of Surgeons Committee on Trauma's Stop the Bleed curriculum. Each participant number will be assigned to each volunteer to maintain anonymity and for accounting purposes.
  Each participant will be isolated and observed by the investigator as he/she attempts to apply a tourniquet to a simulated leg amputation simulator (BCon Trainer, Techline Technologies, Willow Grove, PA). As the participant proceeds with the application of the tourniquet the observer will compare the steps in the tourniquet application process with the steps on data collection form noting any deviations ("YES" for correct, "NO" for deviation or failure to follow that step). Also noted will be total time to complete the tourniquet application process. The raw data from each form will be transferred to a master spread sheet for ease of data analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Somerville EMS Headquarters, Somerville, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
All raw data and methodology will be shared upon study completion
Supporting Information: ICF, CSR
Time Frame: December 2019 through June 30 2019
Access Criteria: email the investigator at sweinman@somervillenj.org